CLINICAL TRIAL: NCT04466449
Title: Different Methods for Detection and Identification of Entamoeba Species in Assuit Governorate Hospitals.
Brief Title: Identification of Entamoeba Spp. in Assuit Governorate Hospitals.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youstina Talaat Basaly, YTalaatBasaly, Assiut University
Other Study IDs: Entamoeba spp. Identification
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Entamoeba Spp. Identification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: stool sample — A stool sample will be collected from each patient for diagnosis of Entamoeba

SUMMARY:
1. Determination the prevalence of Entamoeba histolytica infections among patients at Assiut University Hospitals presented with diarrhea/dysentery.
2. Evaluatation the role of different cultures in diagnosing Entamoeba .
3. Molecularly differentiation between Entamoeba species to monitor the true prevalence of E.histolytica .

DETAILED DESCRIPTION:
Entamoeba histolytica is a common pathogenic protozoan widely distributed throughout the world (10% of the world's population), with 50,000-100,000 deaths reported annually(1) .It is a health problem both in Egypt and worldwide (2) The disease is more prevalent in densely populated areas with poor hygiene requirements and lacking sanitary water supply, especially in rural areas(3). It causes many digestive complications including diarrhea , and fever(2). it transmits through bloodstream forming abscesses in the brain, eye, liver and other vital organs and tissues or even lead to death in some cases . Some individuals have no symptom of the disease but transmit the infection to others(4) It is well- established that E. histolytica leads to invasive disease in humans. Although both E. dispar and E. moshkovskii are still considered to be non pathogenic and free-living amoebas, respectively, some reports suggest their potential role in provoking disease in humans (5) Cysts of E.dispar , E.moshkovskii and E.hartmanni can be confused with E.histolytica. cysts in the parasitological examination(6) The molecular assays, is preferable as it detects E. histolytica , differentiates it from other species and monitors its true prevalence for better treatment and effective control (2)

ELIGIBILITY:
Inclusion Criteria:

* : Male and female patients of different age groups with diarrhea/dysentery attending the outpatient clinics at Assiut University Hospitals .

Exclusion Criteria:

* No exclusion criteria .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients of different age groups with diarrhea/dysentery attending the outpatient clinics at Assiut University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Determination the prevalence of Entamoeba histolytica infections among patients at Assiut University Hospitals presented with diarrhea/dysentery | 2022
  Different Methods for Detection and Identification of Entamoeba species in Assuit Governorate.

CONTACTS AND LOCATIONS:
Locations (1):
- Youstina Talaat, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided